CLINICAL TRIAL: NCT06342206
Title: Attending Physician, Department of Chinese Medicine
Brief Title: The Assessment of Acute /Chronic Phase in Patients With Ischemic Cerebral Stroke Using TCM Diagnostic Tools
Status: Recruiting | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH111-REC2-144
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic
Keywords: stage of stroke, tongue diagnosis, pulse diagnosis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — photography
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral infarction is the second cause of death and the third cause of disability. More than 13.7 million patients worldwide are diagnosed with stroke every year, and the number of deaths is 5.5 million, of which ischemic stroke is the major type, accounting for 87%. Sequelae of stroke are problems that require long-term medical care. If we can intervene and assist with Traditional Chinese Medicine (TCM) at early stage, it will be a great boon for patients. In clinical practice, TCM collects data as the basis for diagnosis through the four diagnostic methods-look, listen, question, and feel the pulse. Among these, tongue diagnosis and pulse diagnosis belong to the categories of look and feel the pulse. At present, the objective examination instruments of TCM developed are mainly tongue diagnostic instruments and pulse diagnostic instruments. Therefore, we hope to utilize tongue and pulse diagnoses as the main reference to analyze the changes in ischemic stroke stages. The data of this study are collected from China Medical University Hospital and YuanRung Hospital-for further statistical analysis. Ischemic stroke patients (ICD-10: I63) who were hospitalized within 1 week from the date of diagnosis were eligible to join this research project. Tongue and pulse examinations were collected once per week within 1 month. A total of 4 tongue-pulse examinations were collected in each case, which were categorized into acute stage (24 hours to 1 week), subacute stage (1 to 3 weeks) and chronic stage (more than 3 weeks). [30] This research is to study the changes of tongue and pulse diagnoses in acute, subacute and chronic stages among ischemic patients who receive TCM diagnosis and treatment. Through utilizing objective evaluation of Chinese and Western medical examination instruments, we hope to establish clear diagnostic standards for TCM syndrome types, so as to evaluate the efficacy of clinical diagnosis and treatment. The goal is to improve the quality of TCM care and to provide Chinese and Western integrated treatment for stroke patients in the future. This research can also serve as a reference for related TCM research and development.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 40 years of age, who acted in concert with the complete examination and answered the questionnaire.
2. Participants were diagnosed as ischemic stroke (ICD-10：I63) by neurologist, and were approved by head CT or MRI examination.
3. Those with a stable vital sign after being examined by an internal medicine specialist
4. Those who experience a cerebral vascular accident within 10 days of the consultation
5. Signing the agreement document to join the research program

Exclusion Criteria:

1. Those with an unstable vital sign
2. Patients who were unable to protrude their tongue or the protruding length was insufficient
3. Those at risk of jaw dislocation
4. Those with an arteriovenous shunt or fistula
5. Those who experience seizures
6. Those with poor cognition and communication

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients in acute phase within 1 week will be included, and continues to collect their data in 2~3 Weeks and 4 week.
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2025-03-27 (Estimated)

PRIMARY OUTCOMES:
Differences between tongue diagnosis and pulse diagnosis in acute and chronic stroke patients | Beginning September 2022 through October 2024
  To compare the differences between tongue and pulse diagnosis in acute, subacute and chronic phases of stroke patients using statistical methods.

CONTACTS AND LOCATIONS:
Locations (1):
- YuanRung Hospital, Changhua, Taiwan